CLINICAL TRIAL: NCT03471923
Title: Non-Motor Features of Cervical Dystonia
Brief Title: Non-Motor Features of Cervical Dystonia (CD)
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mallory Hacker, Research Instructor, Vanderbilt University Medical Center
Other Study IDs: 171717
Record Dates: First submitted 2018-02-23; First posted 2018-03-21 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Cervical Dystonia; Movement Disorders; Focal Dystonia; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations; Neuromuscular Manifestations; Spasmodic Torticollis
MeSH Terms: conditions — Torticollis; Movement Disorders; Dystonic Disorders; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations; Neuromuscular Manifestations | interventions — Neurologic Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CD Patients: Subjects must have a prior diagnosis of cervical dystonia and be capable of participating in all study procedures. Subjects will undergo assessment of non-motor features.
  Interventions: Diagnostic Test: Assessment of Non-Motor Features
- Family Members: Subjects must be a first order relation of a Vanderbilt patient diagnosed with cervical dystonia. The subject must pass a short neurological examination to ensure the subject does not have cervical dystonia or any sensory deficits. Subjects will undergo assessment of non-motor features.
  Interventions: Diagnostic Test: Neurological Examination; Diagnostic Test: Assessment of Non-Motor Features
- Healthy volunteers: Subjects must be healthy volunteers who are neurologically normal. The subject must pass a short neurological examination to ensure the subject does not have cervical dystonia or any sensory deficits. Subjects will undergo assessment of non-motor features.
  Interventions: Diagnostic Test: Neurological Examination; Diagnostic Test: Assessment of Non-Motor Features

INTERVENTIONS:
Diagnostic Test: Neurological Examination — The family members and healthy volunteers will undergo elements of the neurological examination during which the movement disorders neurologist will look specifically for the presence of cervical dystonia and other sensory abnormalities. If the subject is found to have cervical dystonia or any other sensory abnormalities, the subject will be excluded from the study.
  Groups: Family Members; Healthy volunteers
Diagnostic Test: Assessment of Non-Motor Features — All subjects will be assessed for four non-motor symptoms, including (1) spatial discrimination threshold, (2) temporal discrimination threshold, (3) vibration-induced illusion of movement, and (4) kinesthesia.

SUMMARY:
This study will examine the prevalence of four previously identified non-motor markers in a population of cervical dystonia patients, unaffected family members, and healthy volunteers in an attempt to identify a distinct combination of non-motor symptoms that may be indicative of disease development.

DETAILED DESCRIPTION:
The primary aim of this study is to identify the prevalence of four previously identified non-motor markers - (1) spatial discrimination threshold, (2) temporal discrimination threshold, (3) vibration-induced illusion of movement, and (4) kinesthesia - in a population of cervical dystonia patients, unaffected family members, and healthy volunteers (control group). Consenting participants will receive a neurological examination performed by a movement disorders neurologist, followed by an assessment of the four non-motor symptoms.

The investigators hypothesize that a distinct combination of non-motor symptoms will be more prevalent in the CD group, and therefore this set of symptoms may be indicative of disease development. This combination will be identified through analysis of the concurrence of the non-motor features across the three groups of participants. This study will fill an important unmet need, as to the investigators' knowledge there are no published studies assessing the comorbid presentation of these four non-motor symptoms in a single cervical dystonia population. The exploration of a distinct combination of concurrent non-motor symptoms as a marker for the development of cervical dystonia will improve the ability of movement disorders neurologists to diagnose the condition.

The results of this study will facilitate the investigators' longstanding aim of improving rates of cervical dystonia diagnosis. Cervical dystonia is currently diagnosed based upon the exclusion of other movement disorders; therefore, characterization of non-motor features in cervical dystonia patients will help to refine the diagnostic criteria for this condition. This investigation will also improve understanding of the factors associated with CD. Future studies can examine the source of these associated factors in order to help understand the cause of CD, since the etiology is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cervical dystonia, OR a first order relation of a Vanderbilt patient diagnosed with cervical dystonia, OR a healthy volunteer who is neurologically normal
* Capable of participating in all study procedures
* Willing and able to provide written or verbal informed consent.

Exclusion Criteria:

* Subjects for whom participation in the study may cause medical harm
* Subjects who are not considered competent to make their own medical decisions
* Subjects who display sensory deficits during a short screening examination prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will include adults that have cervical dystonia, are healthy and related to someone with cervical dystonia, or are healthy and not related to someone with cervical dystonia (control group).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of spatial discrimination threshold in cervical dystonia patients, unaffected family members, and healthy volunteers | Up to 6 months after consent is obtained
  For participants in all groups, the investigators will examine the prevalence of spatial discrimination threshold. Prevalence of spatial discrimination threshold will be determined with a task using Johnson-Van-Boven-Phillips (JVP) domes. The spatial discrimination threshold will be recorded as the mean of both hands at the 75% level of accuracy. The research coordinator will report prevalence of spatial discrimination threshold as a descriptive statistic.
Prevalence of temporal discrimination threshold in cervical dystonia patients, unaffected family members, and healthy volunteers | Up to 6 months after consent is obtained
  For participants in all groups, the investigators will examine the prevalence of temporal discrimination threshold. Prevalence of temporal discrimination threshold will be determined with a visual-visual discrimination task.The research coordinator will report prevalence of temporal discrimination threshold as a descriptive statistic.
Prevalence of vibration-induced illusion of movement in cervical dystonia patients, unaffected family members, and healthy volunteers | Up to 6 months after consent is obtained
  For participants in all groups, the investigators will examine the prevalence of vibration-induced illusion of movement. Prevalence of vibration-induced illusion of movement will be determined by recording the change in displacement of the tracking arm during a vibration-induced illusion of movement task. The research coordinator will report prevalence of vibration-induced illusion of movement as a descriptive statistic.
Prevalence of impaired kinesthesia in cervical dystonia | Up to 6 months after consent is obtained
  For participants in all groups, the investigators will examine the prevalence of impaired kinesthesia. Kinesthesia will be determined by a neurologist during the neurological examination. The research coordinator will report prevalence of impaired kinesthesia as a descriptive statistic.

SECONDARY OUTCOMES:
Probability of concurrence of multiple non-motor features | Up to 6 months after consent is obtained
  The concurrence of multiple non-motor symptoms will be assessed using a multinomial logistic regression model to determine if a distinct combination of non-motor symptoms is more prevalent in the cervical dystonia patient group than in the unaffected family members or healthy volunteer groups.

OTHER OUTCOMES:
Potential new demographic indicators of cervical dystonia | Up to 6 months after consent is obtained
  Analysis of demographic factors will be performed to identify additional environmental factors that are more prevalent in the CD patient population than in healthy controls and unaffected family members. Through exploration of potential new indicators, the investigators hope to progress the long-term goal of improving the rate of cervical dystonia diagnosis.
Potential new medical indicators of cervical dystonia | Up to 6 months after consent is obtained
  Analysis of medical history and specific elements of the neurological examination will be performed to identify additional symptoms and environmental factors that are more prevalent in the CD patient population than in healthy controls and unaffected family members. Emphasis will be placed on sensory tricks, as previous studies and clinical experience have shown that patients often use sensory tricks such as touching the face, hand, or neck to temporarily relieve muscle contraction. Through exploration of potential new indicators, the investigators hope to progress the long-term goal of improving the rate of cervical dystonia diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowner BE. Cervical dystonia: disease profile and clinical management. Phys Ther. 2007 Nov;87(11):1511-26. doi: 10.2522/ptj.20060272. Epub 2007 Sep 18. PMID 17878433
- [Background] Stacy M. Epidemiology, clinical presentation, and diagnosis of cervical dystonia. Neurol Clin. 2008 May;26 Suppl 1:23-42. doi: 10.1016/s0733-8619(08)80003-5. No abstract available. PMID 18603166
- [Background] Jinnah HA, Berardelli A, Comella C, Defazio G, Delong MR, Factor S, Galpern WR, Hallett M, Ludlow CL, Perlmutter JS, Rosen AR; Dystonia Coalition Investigators. The focal dystonias: current views and challenges for future research. Mov Disord. 2013 Jun 15;28(7):926-43. doi: 10.1002/mds.25567. PMID 23893450
- [Background] Stamelou M, Edwards MJ, Hallett M, Bhatia KP. The non-motor syndrome of primary dystonia: clinical and pathophysiological implications. Brain. 2012 Jun;135(Pt 6):1668-81. doi: 10.1093/brain/awr224. Epub 2011 Sep 20. PMID 21933808
- [Background] Bradley D, Whelan R, Kimmich O, O'Riordan S, Mulrooney N, Brady P, Walsh R, Reilly RB, Hutchinson S, Molloy F, Hutchinson M. Temporal discrimination thresholds in adult-onset primary torsion dystonia: an analysis by task type and by dystonia phenotype. J Neurol. 2012 Jan;259(1):77-82. doi: 10.1007/s00415-011-6125-7. Epub 2011 Jun 8. PMID 21656045
- [Background] Chen H, Zhao EJ, Zhang W, Lu Y, Liu R, Huang X, Ciesielski-Jones AJ, Justice MA, Cousins DS, Peddada S. Meta-analyses on prevalence of selected Parkinson's nonmotor symptoms before and after diagnosis. Transl Neurodegener. 2015 Jan 8;4(1):1. doi: 10.1186/2047-9158-4-1. eCollection 2015. PMID 25671103
- [Background] Frima N, Nasir J, Grunewald RA. Abnormal vibration-induced illusion of movement in idiopathic focal dystonia: an endophenotypic marker? Mov Disord. 2008 Feb 15;23(3):373-7. doi: 10.1002/mds.21838. PMID 18044715
- [Background] Molloy FM, Carr TD, Zeuner KE, Dambrosia JM, Hallett M. Abnormalities of spatial discrimination in focal and generalized dystonia. Brain. 2003 Oct;126(Pt 10):2175-82. doi: 10.1093/brain/awg219. Epub 2003 Jun 23. PMID 12821512
- [Background] Fiorio M, Gambarin M, Valente EM, Liberini P, Loi M, Cossu G, Moretto G, Bhatia KP, Defazio G, Aglioti SM, Fiaschi A, Tinazzi M. Defective temporal processing of sensory stimuli in DYT1 mutation carriers: a new endophenotype of dystonia? Brain. 2007 Jan;130(Pt 1):134-42. doi: 10.1093/brain/awl283. Epub 2006 Nov 14. PMID 17105745
- [Background] Bradley D, Whelan R, Walsh R, O'Dwyer J, Reilly R, Hutchinson S, Molloy F, Hutchinson M. Comparing endophenotypes in adult-onset primary torsion dystonia. Mov Disord. 2010 Jan 15;25(1):84-90. doi: 10.1002/mds.22889. PMID 19938165
- [Background] Westenberger A, Klein C. Genetics of dystonia. In: Dystonia and Dystonic Syndromes. ; 2015:27-48. doi:10.1007/978-3-7091-1516-9_3.
- [Background] Putzki N, Stude P, Konczak J, Graf K, Diener HC, Maschke M. Kinesthesia is impaired in focal dystonia. Mov Disord. 2006 Jun;21(6):754-60. doi: 10.1002/mds.20799. PMID 16482525
- [Background] Walsh R, O'Dwyer JP, Sheikh IH, O'Riordan S, Lynch T, Hutchinson M. Sporadic adult onset dystonia: sensory abnormalities as an endophenotype in unaffected relatives. J Neurol Neurosurg Psychiatry. 2007 Sep;78(9):980-3. doi: 10.1136/jnnp.2006.105585. PMID 17702779
- [Background] Bradley D, Whelan R, Walsh R, Reilly RB, Hutchinson S, Molloy F, Hutchinson M. Temporal discrimination threshold: VBM evidence for an endophenotype in adult onset primary torsion dystonia. Brain. 2009 Sep;132(Pt 9):2327-35. doi: 10.1093/brain/awp156. Epub 2009 Jun 12. PMID 19525326
- [Background] Klingelhoefer L, Martino D, Martinez-Martin P, et al. Nonmotor symptoms and focal cervical dystonia: Observations from 102 patients. Basal Ganglia. 2014;4(3-4):117-120. doi:10.1016/j.baga.2014.10.002.
- [Background] Lobbezoo F, Tanguay R, Thon MT, Lavigne GJ. Pain perception in idiopathic cervical dystonia (spasmodic torticollis). Pain. 1996 Oct;67(2-3):483-91. doi: 10.1016/0304-3959(96)03153-3. PMID 8951945
- [Background] Defazio G, Jankovic J, Giel JL, Papapetropoulos S. Descriptive epidemiology of cervical dystonia. Tremor Other Hyperkinet Mov (N Y). 2013 Nov 4;3:tre-03-193-4374-2. doi: 10.7916/D80C4TGJ. eCollection 2013. PMID 24255801